CLINICAL TRIAL: NCT06436560
Title: Support for Transgender and Non-Binary Individuals Seeking Vaginoplasty (STRIVE) Study
Brief Title: Support for Transgender and Non-Binary Individuals Seeking Vaginoplasty Study
Acronym: STRIVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); NYU Langone Health (Other); Rush University (Other); University of Utah (Other); University of Minnesota (Other); Temple University (Other); University of California, San Francisco (Other); University of Washington (Other); Trans Lifeline (Unknown); Whitman-Walker Institute (Other Government); Duke University (Other)
Responsible Party: Principal Investigator, Geolani Dy, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00026957; 1023677 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Gender Affirmation Surgery; Perioperative Care; Transgender Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STRIVE Peer Support Intervention (Experimental): A virtual group-based peer support intervention led by trans peers who have had genital gender-affirming surgery.
  Interventions: Other: STRIVE Peer Support Intervention
- Enhanced Usual Care (No Intervention): Usual care enhanced with written and web-based education materials.

INTERVENTIONS:
Other: STRIVE Peer Support Intervention — A virtual group-based peer support intervention led by trans peers who have had genital gender-affirming surgery.
  Arms: STRIVE Peer Support Intervention

SUMMARY:
The STRIVE study is the first national randomized trial to focus on improving well-being, access to surgical care and other health outcomes for transgender and nonbinary (referred to as trans) people seeking genital gender-affirming surgery (GGAS). Trans people have gender identities that are different from the sex they were assigned at birth. Due to discrimination based on their gender identity in settings such as schools, the workplace, housing and health care, trans people face much higher rates of distress as well as poorer health and quality of life. Trans people are often unable to access necessary surgeries and hormone therapy to help align their bodies with their gender identities due to a lack of trained medical providers and limited insurance coverage for gender-affirming care.

The most common GGAS that trans people seek is vaginoplasty, which is the surgical creation of vaginal anatomy. Because of the high demand for this surgery and limited number of medical centers that offer it, trans people face lengthy wait times and complicated health system processes, increasing stress, negative mental health effects and social isolation. Social and peer-support interventions have been shown to decrease isolation and improve health. Social support during the GGAS process was also identified by the Transgender and Non-Binary Surgery - Allied Research Collective (TRANS-ARC) as the top research priority. Due to limited information on this topic, the STRIVE study was developed to meet this need.

The research team's goals are to:

* Compare the effectiveness of two approaches to presurgical preparation for vaginoplasty: a virtual group-based peer support intervention led by trans peers who have had GGAS, or usual care delivered by gender-affirming surgical teams, enhanced with patient education materials.
* Determine if the intervention improves meeting presurgical criteria for vaginoplasty.
* Evaluate if patients, peer supporters and healthcare staff find the intervention acceptable.

The research team will conduct a pragmatic randomized controlled trial, meaning participants will be assigned by chance to one of two groups: peer-support group or usual care enhanced with written and web-based education materials. This study is pragmatic because it is happening under real-life conditions to understand if the intervention will work in practice.

The research team will work with five academic gender-affirming surgery programs across the country to recruit and enroll 260 trans adults ages 18 and older who are seeking vaginoplasty. Participants assigned to the peer support group will receive the intervention virtually over the course of three months, facilitated by peer facilitators from Trans Lifeline. The usual care group will receive education from their gender-affirming surgical team, with in-depth materials that cover the same topics as the virtual course.

The primary outcome to be measures at six months is coping self-efficacy, reported by patients, using a survey which assesses perceived ability to deal with stressors. The research team will explore additional outcomes at 12 months, including meeting GGAS presurgical criteria and other outcomes deemed important to trans community partners, surgeons and other gender-affirming providers (e.g., psychological stress, social support, resilience, quality of life, presurgical knowledge, surgical delays and cancellations). Postsurgical outcomes, including surgical satisfaction and other related outcomes, will be measured at 24 months. Finally, the team will conduct in-depth interviews with participants who undergo the intervention to understand their experiences at the beginning of the study and after six months. Researchers will also interview peer supporters and clinicians to understand how to improve and implement the support intervention more broadly.

In designing this study, the research team worked closely with trans community members and patients, health services and policy researchers, gender-affirming surgeons, advocates, gender program administrators and representatives from social support organizations. Collaboration with and input from the trans community during the conduct of this study will be critical to ensure that the STRIVE study is patient centered. Results from this study will be shared in multiple forms, including clinical guideline recommendations, policy briefs, patient-centered reports, web-based information and summaries for clinicians and researchers. Trans people seeking gender-affirming surgery can use the study findings to understand options for social support to improve quality of life and health outcomes. Clinicians, gender program administrators, health insurance companies and health policy advisors can use the findings from this study to better support and prepare patients who are seeking gender-affirming surgery.

DETAILED DESCRIPTION:
OUTLINE The STRIVE (Support for Transgender and Non-Binary Individuals Seeking Vaginoplasty) Study is a multi-site, two-arm randomized pragmatic trial to determine if an evidence-based peer support intervention improves patient-reported and patient-centered clinical outcomes for individuals seeking genital gender-affirming surgery (GGAS) compared with enhanced usual care.

PRIMARY OBJECTIVES Aim 1: To compare the effectiveness of a virtual, group-based perioperative peer support intervention with enhanced usual care on coping self-efficacy (primary outcome) among patients seeking vaginoplasty.

* Hypothesis 1: Patients in the intervention arm will have greater improvements in coping self-efficacy at 6 months post-enrollment compared to patients who receive enhanced usual care.

Aim 2: To determine whether our perioperative peer support intervention improves patient probability of meeting pre-operative GGAS criteria (secondary outcome), and other prioritized patient-centered outcomes (exploratory outcomes).

* Hypothesis 2a: More patients in the intervention arm will meet pre-operative GGAS criteria at 12 months post-enrollment compared with patients who receive enhanced usual care.
* Hypotheses 2b: Patients in the intervention arm will have decreased psychological distress (anxiety, depression, suicidal ideation) and gender minority stress, and greater social support, resilience, QOL, pre-operative surgical knowledge, and fewer surgical delays. For participants who undergo surgery during the follow-up period, those in the intervention arm will have fewer surgical complications, greater completion of vaginal dilation, greater surgical satisfaction, and fewer unplanned emergency department and clinic visits at 6 months post-operatively.

Aim 3: To evaluate the acceptability of this centralized, virtual, group-based perioperative peer support intervention among patients, peer support specialists and healthcare team members.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified trans or non-binary individual
* Seeking vaginoplasty
* Completed consultation with gender-affirming surgeon for vaginoplasty
* Documented recommendation by surgeon for vaginoplasty
* Can complete survey responses online, by phone or on paper.
* Willing and able to participate in virtual peer support intervention
* Aged 18 or older
* English speaking
* Able to provide independent written consent

Exclusion Criteria:

* Do not speak English
* Cannot complete survey responses online, by phone, or on paper
* Are unwilling to participate in a virtual peer support intervention
* Have co-morbidities or other conditions that exclude them from candidacy for vaginoplasty
* Are currently involved in delivery of the STRIVE Intervention
* Are unable or unwilling to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender and nonbinary persons seeking gender-affirming vaginoplasty.
Enrollment: 260 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-reported coping self-efficacy as assessed by the CSES | Enrollment, 6 months after enrollment, 6 months post-operative
  Patient-reported coping self-efficacy is measured using the Coping Self-Efficacy Scale (CSES), a survey that assesses the perceived ability to deal with stressors using a score range of 0-260. Zero is equivalent to no perceived ability to deal with stressors; 260 indicates the highest attainable level of perceived ability to deal with stressors.

SECONDARY OUTCOMES:
Completion of preoperative criteria for scheduling GGAS | Enrollment, 12 months after enrollment
  Completion of pre-operative criteria for scheduling genital gender-affirming surgery (GGAS), a proxy for patient readiness that is assessed based on each patient's ability to meet criteria of the center at which they are seeking care. Pre-operative criteria generally follow the World Professional Association for Transgender Health (WPATH) Standards of Care (SOC), which have been adopted by most public and private insurers in making coverage decisions for GGAS. WPATH SOC criteria include: a letter of support from a mental health professional attesting to one's ability to provide informed consent stability of ones' gender identity and desire for surgery, and that any mental health and/or medical conditions are well-managed. Additional center-specific requirements may also include: meeting weight criteria; nicotine cessation; glycemic control; and attestation of adequate social support and post-operative housing stability.

OTHER OUTCOMES:
Health-related quality of life assessed by the PROMIS-29 Profile v2.0 | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 Profile v2.0. PROMIS tools were developed to be disease non-specific measures of health-related domains such as self-efficacy for symptom and medication management, depression, anxiety, fatigue, pain interference, sleep disturbance, and physical functioning. Each domain in composed of an item bank specific to a trait being measured. Item banks are calibrated on a common scale to facilitate comparability across varying populations. Raw scores are transformed to standardized T-score metrics, with a mean of 50 and standard deviation of 10.
Depression assessed by the PHQ-9 | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The Patient Depression Questionnaire-9 (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. The PHQ-9 incorporates the Diagnostic and Statistical Manual of Mental Disorders (DSM) depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The score ranges from zero to 27, with zero representing no depression and 27 representing severe depression.
Anxiety assessed by the GAD-7 | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The Generalised Anxiety Disorder Assessment (GAD-7) is a seven-item instrument that is used to measure or assess the severity of generalized anxiety disorder (GAD). Scores range from zero, representing minimal anxiety, to 21, representing severe anxiety.
Presurgical GGAS knowledge assessed by the GENDER-Q "Information" scale | Enrollment, 6 months after enrollment, immediate pre-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Information" scale of the GENDER-Q assesses patient satisfaction with presurgical genital gender-affirming surgery (GGAS) knowledge. Scores range from 27 to 135, with 27 representing not at all satisfied and 135 representing extremely satisfied.
Complications and adverse effects assessed by the GENDER-Q "Adverse Effects" scale | Immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Adverse Effects" scale of the GENDER-Q assesses patient concerns about ongoing problems caused by gender-affirming surgery. Scores range from 30 to 150, with 30 representing not at all concerned and 150 representing extremely concerned.
Gender dysphoria life impact assessed by the GENDER-Q "Gender dysphoria life impact" scale | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. Gender dysphoria describes a state of discomfort or distress a person can experience when their gender identity differs from their sex assigned at birth. The "Gender dysphoria life impact" scale of the GENDER-Q assesses how often gender dysphoria negatively interferes with the patient's life. Scores range from 16 to 80, with 16 representing gender dysphoria never negatively interferes and 80 representing gender dysphoria always negatively interferes.
Social support assessed by the MSPSS | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The Multi-Dimensional Scale of Perceived Social Support (MSPSS) is a 12-item measure of perceived adequacy of social support from three sources: family, friends, and significant other, using a 5-point Likert scale (0 = strongly disagree, 5 = strongly agree). To calculate mean scores, sum across all 12 items, then divide by 12. Scores ranging from 1 to 2.9 are low support; a score of 3 to 5 is moderate support; a score from 5.1 to 7 is considered high support.
Sexual function assessed by the GENDER-Q "Sexual well-being" scale | Enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Sexual well-being" scale of the GENDER-Q assesses satisfaction with sexual activities. Scores range from 16 to 80, with 16 representing never satisfied with sexual activities and 80 always satisfied with sexual activities.
Bodily appearance satisfaction assessed by the GENDER-Q "Appearance" scale | Enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Appearance" scale of the GENDER-Q assesses satisfaction with appearance in relation to gender identity. Scores range from 14 to 70, with 14 representing never satisfied with appearance and 70 always satisfied with appearance.
Urinary function assessed by the GENDER-Q "Urinary function" scale | Immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Appearance" scale of the GENDER-Q assesses satisfaction with appearance in relation to gender identity. Scores range from 14 to 70, with 14 representing never satisfied with appearance and 70 always satisfied with appearance.
Satisfaction with healthcare team assessed by the GENDER-Q "Healthcare professional" and "Gender clinic" scales | Enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The"Healthcare professional" and "Gender clinic" scales of the GENDER-Q assess the patient's satisfaction with the healthcare team providing gender-affirming care. Scores range from 54 to 324, with 54 representing very unsatisfied with the healthcare team and 324 representing completely satisfied with the healthcare team.
Satisfaction with vagina assessed by the GENDER-Q "Vagina" scale | Immediate post-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Vagina" scale of the GENDER-Q assesses satisfaction with the patient's vagina after gender-affirming vaginoplasty. Scores range from 22 to 132, with 22 representing extremely dissatisfied and 132 representing extremely satisfied.
Satisfaction with surgical outcome assessed by the GENDER-Q "Outcome of surgery" scale | Immediate post-operative, 3 months post-operative, 6 months post-operative
  The GENDER-Q is a comprehensive patient-reported outcome measure used to evaluate outcomes of psychological, hormonal, and surgical gender-affirming treatments. The "Outcome of surgery" scale of the GENDER-Q assesses the patient's overall satisfaction with the gender-affirming surgery. Scores range from 17 to 102, with 17 representing extremely dissatisfied and 102 representing extremely satisfied.
Gender minority stress and resilience assessed by the GMSR | Enrollment, 6 months after enrollment, immediate pre-operative, 3 months post-operative, 6 months post-operative
  The Gender Minority Stress and Resilience (GMSR) measure was developed to assess aspects of minority stress and resilience faced by people whose gender identity or expression is different in any way from that socially expected based on their sex assigned at birth. The measure is scored in three subscales. For distal stressors (e.g., gender-related discrimination), scores range from zero, indicating no experience of distal minority stressors, to 60, indicating the greatest degree of experience of distal stressors. For proximal stressors (e.g., internalized transphobia), scores range from zero, indicating no experience of proximal minority stressors, to 88, indicating the greatest degree of experience of proximal stressors. For resilience factors (e.g., community connectedness), scores range from zero, indicating no resilience factors, to 52, indicating the greatest degree of resilience factors.

CONTACTS AND LOCATIONS:
Overall Officials: Geolani Dy, MD, Principal Investigator — Oregon Health and Science University
Locations (8):
- United States (8):
  - University of California San Francisco, San Francisco, California
  - Rush University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - New York University Langone Health, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Temple University, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Due to safety concerns about the use of data expressed during patient engagement processes, the STRIVE Study does not currently plan to share individual participant data (IPD) publicly.